CLINICAL TRIAL: NCT01863875
Title: Assessment of Listening, Speech, and Language Proficiency, and of Experienced Quality of Life in People Who Have Received Cochlear Implants as Children.
Brief Title: Language Proficiency and Quality of Life After Receiving Cochlear Implantation as a Child
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Oslo University Hospital (Other)
Collaborators: University of Oslo (Other); Norwegian Directorate of Health (Other Government)
Responsible Party: Principal Investigator, Ona Bø Wie, Professor, Oslo University Hospital
Other Study IDs: 2012/2154
Record Dates: First submitted 2013-05-23; First posted 2013-05-29 (Estimated); Last update posted 2016-04-07 (Estimated); Status verified 2016-04

CONDITIONS: Hearing Loss
Keywords: Cochlear Implant; Hearing loss; Language Development; Quality of life
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Childhood cochlear implant recipients: The sample includes all childhood cochlear implant (CI) recipients at Oslo University Hospital in Norway from 1988-2012. The participant must have at least one year of CI-user time. Possible sample size is 530 children. The age span is from 1 to 50 years.
- Normal hearing people: Reference group: A group of normal hearing people matching the target group on gender and age.

SUMMARY:
Treatment with cochlear implantation is now offered to proximately 95 % of children with deafness in Norway. More than 500 children have been operated at Oslo University Hospital. The study is a cross-sectional study aimed to investigate speech perception, language skills, quality of life in all childhood cochlear implant (CI) recipients in Norway from 1988-2012. Factors such as child characteristics, characteristics with the family, the cochlear implant, the rehabilitation situation, choice of communication mode, school and work situation are surveyed to see if these factors can be associated with variations in outcome. The study will include pre and post lingual deaf children and children with multiple disabilities. Participants are recruited and examined in conjunction with their annual CI control at the hospital. It will be conducted a series of tests determining listening, speech and language development, non-verbal intelligence. Questionnaires are used to collect background information and quality of life experience. The questionnaires include self-report forms for different age groups, and a parent report form. The patient will be tested for the most common genetic causes of deafness. Additional data will be collected from patient records and from local health register at Oslo University Hospital.

DETAILED DESCRIPTION:
Test protocol includes:

Hearing and Language assessment:

Single syllable word perception, Hearing in noise test (HINT), Mullen Scale of Early Learning, British Picture Vocabulary Scale, Peabody Picture Vocabulary Test - Fourth Edition, Clinical Evaluation of Language Fundamentals (CELF) - Fourth Edition 4 , Raven progressive matrices, Motor Coordination + Visual Perception (VMI), Wechsler Preschool and Primary Scale of Intelligence (WPPSI), Wechsler Intelligence Scale for Children (WISC) and Wechsler Adult Intelligence Scale (WAIS).

Quality of Life assessment:

Satisfaction of Life Scale for Children Pediatric Quality of Life Inventory TM (PedsQL TM) Questionnaire for quality of life assessments (KINDL)

ELIGIBILITY:
Inclusion Criteria:

* All people in Norway that have received Cochlear implants as a child and that have one or more than one year with CI experience.

Exclusion Criteria:

* Cochlear implant users with less than one year with CI experience and people implanted after 18 years of age.

Ages: 18 Months to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All people in Norway that have received Cochlear Implants as a child.
Sampling Method: Non-Probability Sample
Enrollment: 530 (Estimated)
Dates: Start 2013-01; Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Hearing and listen skills | 2013-2023 (up to 20 years)
  Single syllable word perception, HINT hearing in noise test

SECONDARY OUTCOMES:
Speech and language skills | 2013-2032 (up to 20 years)
  Mullen Scale of Early Learning, British Picture Vocabulary Scale Clinical Evaluation of Language Fundamentals - Fourth Edition 4 CELF

OTHER OUTCOMES:
Quality of life | 2013-2023 (up to 20 years)

CONTACTS AND LOCATIONS:
Overall Officials: Terje A Osnes, Professor, Study Chair — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Department of Otolaryngology, Olso, Olso, Norway

IPD SHARING:
Plan to Share IPD: No